CLINICAL TRIAL: NCT04574089
Title: Medical Ethics Committee of Peking University Shenzhen Hospital
Brief Title: Treatment for Aerobic Vaginitis by Using Bofukang Vaginal Suppository
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Shangrong Fan, Principal Investigator, Peking University Shenzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUShenzhenH
Record Dates: First submitted 2020-02-20; First posted 2020-10-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Vaginitis
Keywords: Aerobic vaginitis; Treatment
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baofukang Suppository 7 days (Experimental): Baofukang Suppository (1.74g), for vaginal external use, 2 capsules per night for 7 days
  Interventions: Drug: Experimental: Baofukang Suppository 7 days
- Baofukang Suppository 14 days (Experimental): Baofukang Suppository (1.74g), for vaginal external use, 2 capsules per night for 14days
  Interventions: Drug: Experimental: Baofukang Suppository 14 days

INTERVENTIONS:
Drug: Experimental: Baofukang Suppository 7 days — Experimental: Baofukang Suppository 7 days
  Other Names: Baofukang Suppository 7 days
  Arms: Baofukang Suppository 7 days
Drug: Experimental: Baofukang Suppository 14 days — Experimental: Baofukang Suppository 14 days
  Other Names: Baofukang Suppository 14 days
  Arms: Baofukang Suppository 14 days

SUMMARY:
Aerobic vaginitis was treated by using Baofukang Suppository 7 days group or Baofukang Suppository 14 days group.To evaluate the efficacy and safety after treatment.

DETAILED DESCRIPTION:
Aerobic vaginitis was treated by using Baofukang Suppository 7 days group or Baofukang Suppository 14 days group.

Group 1: Baofukang Suppository (1.74g), for vaginal use, 2 capsules per night for 7 days.

Group 2: Baofukang Suppository (1.74g), for vaginal use, 2 capsules per night for 14 days.

The efficacy and safety will be evaluated 7~14 days after treatment and 35~42 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

Aerobic vaginitis diagnosed based on present ：

1. Vaginal dischareg ;
2. pH > 4.5;
3. Donders score≥3;

Exclusion Criteria:

1. Patients with other vaginitis, cervical erosion, or suspected gonorrhea, herpes simplex virus infection and other vulvar diseases;
2. Patients received systemic or vaginal antifungal or antibiotic treatment within two weeks before admission.
3. Pregnancy, lactation and intentional pregnancy;
4. Women with liver and kidney dysfunction, low immune function, diabetes, psychosis or other serious diseases;
5. Allergic constitution and patients allergic to drug ingredients in this study;
6. Those with poor compliance.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with sexual activity
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cure rate | First week after treatment
  A vaginal smear composite Donders score of 1 to 2 represents normality. A score of more than 2 is aerobic vaginitis. There are four variables(Lactobacillary; leucocytes; toxic leukocytes; parabasal cells; background flora). Detail see references Links.
Cure rate | First month after the treatment
  A vaginal smear composite Donders score of 1 to 2 represents normality. A score of more than 2 is aerobic vaginitis. There are four variables(Lactobacillary; leucocytes; toxic leukocytes; parabasal cells; background flora).Detail see folowing references.

SECONDARY OUTCOMES:
Side affect | First week after treatment
  Number of Participants Experiencing AEs Following the First Dose of the Study Product

CONTACTS AND LOCATIONS:
Overall Officials: Shangrong Fan, M.D., Principal Investigator — Dept of Obstetrics and Gynecology,Peking University Shenzhen Hospital
Locations (1):
- Peking University Shenzhen Hosptal, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AV diagnosis and outcome Measure — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8775230/pdf/diagnostics-12-00185.pdf